CLINICAL TRIAL: NCT01173432
Title: Randomized Controlled Trial of the Effect of Continuous Positive Airway Pressure on Adipocyte Fatty Acid Binding Protein and Other Metabolic Markers in Obstructive Sleep Apnea
Brief Title: Exploring the Role of Adipocyte Fatty Acid Binding Protein in the Association of Obstructive Sleep Apnea and Metabolic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Professor Mary SM Ip, The University of Hong Kong, Queen Mary Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW07-178; HKCTR-770 (Registry Identifier: Clinical trial centre, The University of Hong Kong)
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea; Insulin Resistance; Metabolic Syndrome; Inflammation
Keywords: obstructive sleep apnea; metabolic dysfunction; metabolic syndrome; adipocyte fatty acid binding protein
MeSH Terms: conditions — Sleep Apnea, Obstructive; Insulin Resistance; Metabolic Syndrome; Inflammation | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- continuous positive airway pressure (Active Comparator): using continuous positive airway pressure (CPAP) device during sleep, for the study period (4 weeks)
  Interventions: Device: continuous positive airway pressure
- control (No Intervention): observation for the study period (4 weeks, no CPAP)

INTERVENTIONS:
Device: continuous positive airway pressure — an device to be used during sleep, which was a nasal mask connected to a device with pressure applied to upper airway
  Arms: continuous positive airway pressure

SUMMARY:
Adipocyte fatty acid binding protein (A-FABP) is a member of the FABP super family, is abundant in adipocytes and macrophages. Regulatory functions of A-FABP in lipid and glucose metabolism have been described, and it is suggested to play an important role in the pathogenesis of metabolic syndrome.We hypothesize that obstructive sleep apnea (OSA) may upregulate A-FABP production and thus causally contribute to metabolic dysfunction. Our group has recently demonstrated that A-FABP, expressed and secreted from adipocytes, is present in the blood stream .The levels of A-FABP correlated with various metabolic variates in the metabolic syndrome. Furthermore, we have obtained novel data in men with a range of sleep disordered breathing showed that the duration of oxygen desaturation correlated with circulating levels of A-FABP, independent of age and waist/body mass index. The current proposal aims to pursue this finding and further explore the role of A-FABP in the association of OSA and metabolic dysfunction.

DETAILED DESCRIPTION:
We hypothesize that there are changes in circulating A-FABP level which can be mitigated by effective treatment of OSA.

The aim is to investigate the effect of CPAP treatment of OSA on circulating A-FABP, and other metabolic biomarkers and cardiovascular parameters

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 - 65 years old
* Able to understand and give informed written consent

Exclusion Criteria:

* BMI > 35 kg/m2, and features of obesity hypoventilation syndrome
* known diabetes mellitus or hyperlipidemia on treatment
* known cardiovascular disease except hypertension stable on treatment
* unstable medical illness
* need for starting treatment for OSA or other medical conditions immediately

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
adipocyte fatty acid binding protein | changes over 4 weeks of CPAP treatment
  blood assay

SECONDARY OUTCOMES:
Insulin and glucose | changes over 4 weeks of CPAP treatment
  blood assay
Lipids and lipoprotein | changes over 4 weeks of CPAP treatment
  blood assay
blood Markers of oxidative stress and fat metabolism | changes over 4 weeks of CPAP treatment
blood inflammatory markers | changes over 4 weeks of CPAP treatment
blood pressure | changes over 4 weeks of CPAP treatment
Epworth sleepiness scale | changes over 4 weeks of CPAP treatment
  by sleep questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mary SM Ip, MD, Principal Investigator — The University of Hong Kong, Queen Mary Hospital
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Xu A, Wang Y, Xu JY, Stejskal D, Tam S, Zhang J, Wat NM, Wong WK, Lam KS. Adipocyte fatty acid-binding protein is a plasma biomarker closely associated with obesity and metabolic syndrome. Clin Chem. 2006 Mar;52(3):405-13. doi: 10.1373/clinchem.2005.062463. Epub 2006 Jan 19. PMID 16423904
- [Background] Stejskal D, Karpisek M. Adipocyte fatty acid binding protein in a Caucasian population: a new marker of metabolic syndrome? Eur J Clin Invest. 2006 Sep;36(9):621-5. doi: 10.1111/j.1365-2362.2006.01696.x. PMID 16919044
- [Background] Lam DC, Xu A, Lam KS, Lam B, Lam JC, Lui MM, Ip MS. Serum adipocyte-fatty acid binding protein level is elevated in severe OSA and correlates with insulin resistance. Eur Respir J. 2009 Feb;33(2):346-51. doi: 10.1183/09031936.50075408. PMID 19181913
- [Derived] Lui MMS, Mak JCW, Chong PWC, Lam DCL, Ip MSM. Circulating adipocyte fatty acid-binding protein is reduced by continuous positive airway pressure treatment for obstructive sleep apnea-a randomized controlled study. Sleep Breath. 2020 Sep;24(3):817-824. doi: 10.1007/s11325-019-01893-5. Epub 2019 Aug 1. PMID 31372823